CLINICAL TRIAL: NCT01716494
Title: Severe Asthma Research Program (SARP)-Washington University
Brief Title: Washington University Severe Asthma Research Program III
Acronym: WU SARPIII
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201206102
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, DNA, RNA, sputum, urine, bronchial tissue, bronchoalveolar lavage, bronchial brushings, exhaled breath condensate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Severe Asthma: Subjects with severe asthma (SARP protocol definition)
- Well controlled asthma: Subjects with well controlled asthma
- Normal control: Subjects that are healthy normals

SUMMARY:
The overall goal of this proposal is to better understand the basis of airway remodeling in severe asthma and how remodeling changes over time. The investigators propose to study a well-characterized cohort of adult and pediatric subjects with severe asthma using a multidisciplinary state-of-the-art approach.

DETAILED DESCRIPTION:
The overall goal of this proposal is to better understand the molecular basis and structural and physiologic consequences of airway remodeling in severe asthma and how remodeling changes over time. In that context, the investigators propose to study a well-characterized cohort of adult and pediatric subjects with severe asthma using a multidisciplinary approach that includes state-of-the-art morphometric, imaging, and physiologic measurements of airways. The investigators will contrast these findings to those in groups with well-controlled asthma, normal controls, and diseased controls (chronic bronchitis) to identify features that can provide biologic targets unique to severe asthma. The investigators have demonstrated that epithelial hyperplasia, goblet cell metaplasia and mucin production are features of airway remodeling in subjects with severe asthma, and that epithelial remodeling was due to increased epithelial proliferation and decreased cell death. The investigators propose that individuals with severe asthma, in comparison to well controlled asthma, have: (I) increased airway remodeling as evidenced by goblet cell metaplasia and mucin production, (II) greater airway thickness by multidetector-row CT of the chest (MDCT) leading to ventilation defects demonstrated by hyperpolarized helium (3He) MRI and air trapping demonstrated by MDCT, and (III) airway remodeling associated with more severe and progressive airflow obstruction. The investigators hypothesize that the goblet cell metaplasia and increased mucin The investigators have observed in severe asthma are being driven by an IL-13- and EGFR-dependent mechanism that inhibits epithelial cell apoptosis and allows IL-13 differentiation of the airway epithelium into goblet cells (Aim I). The investigators further hypothesize that this remodeling of segmental airways in severe asthma leads to distal ventilation defects and air trapping (Aim II). In an effort to define potential predictors of subsequent decline in lung function in severe asthma, the investigators hypothesize that baseline airway remodeling as reflected by MDCT airway wall area (AWA%) is predictive of FEV1 (post-corticosteroid/bronchodilator FEV1) decline (Aim III). The identification of potential variables associated with remodeling and severe asthma will help identify individuals at risk whom would benefit from specific targeted therapy. The concerted efforts of this project together with the SARP will lead to new insights on the mechanistic basis for severe asthma, further elucidate how it differs from mild-moderate asthma, identify potential targets for intervention, and will provide imaging metrics to objectively evaluate outcomes for new treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosis of asthma,
2. Age 6 years and older
3. Evidence of historical reversibility, including either:

   1. FEV1 bronchodilator reversibility ≥ 12%, or
   2. Airway hyperresponsiveness reflected by a methacholine PC20 ≤16 mg/mL.

Exclusion Criteria:

1. No primary medical caregiver,
2. Pregnancy (if undergoing methacholine challenge or bronchoscopy),
3. Current smoking
4. Smoking history > 10 pack years if ≥ 30 years of age or smoking history > 5 pack years if < 30 years of age (Note: If a subject has a smoking history, no smoking within the past year)
5. Other chronic pulmonary disorders associated with asthma-like symptoms,including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction that is the sole cause of asthma symptoms, severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways,
6. History of premature birth before 35 weeks gestation,
7. Evidence that the participant or family may be unreliable or poorly adherent to their asthma treatment or study procedures,
8. Planning to relocate from the clinical center area before study completion, or
9. Any other criteria that place the subject at unnecessary risk according to the judgment of the Principal Investigator and/or attending physician(s) of record.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with asthma (severe asthma, well controlled asthma) and healthy normal controls from St. Louis region
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Lung function | 3 yrs
  decline in lung function (FEV1) over 3 yrs

SECONDARY OUTCOMES:
Asthma Control Questionnaire | 3 yrs
  asthma control score (ACQ)
Health care utilization | 3 yrs
  Health care utilization including ED visits and hospitalizations.
Exacerbation | 3 yrs
  Exacerbations requiring systemic steroids
CT quantification | 3 yrs
  CT airway wall thickness, lung density
MRI | 3 yrs
  Ventilation defects on hyperpolarized gas MRI
Morphometric biopsy | 3 yrs
  Morphometric analysis of airway biopsies
Gene expression | 3 yrs
  Gene expression studies of airway epithelial cells

CONTACTS AND LOCATIONS:
Overall Officials: Kaharu Sumino, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Huang BK, Elicker BM, Henry TS, Kallianos KG, Hahn LD, Tang M, Heng F, McCulloch CE, Bhakta NR, Majumdar S, Choi J, Denlinger LC, Fain SB, Hastie AT, Hoffman EA, Israel E, Jarjour NN, Levy BD, Mauger DT, Sumino K, Wenzel SE, Castro M, Woodruff PG, Fahy JV, Sarp FTNSARP. Persistent mucus plugs in proximal airways are consequential for airflow limitation in asthma. JCI Insight. 2024 Feb 8;9(3):e174124. doi: 10.1172/jci.insight.174124. PMID 38127464
- [Derived] Dunican EM, Elicker BM, Gierada DS, Nagle SK, Schiebler ML, Newell JD, Raymond WW, Lachowicz-Scroggins ME, Di Maio S, Hoffman EA, Castro M, Fain SB, Jarjour NN, Israel E, Levy BD, Erzurum SC, Wenzel SE, Meyers DA, Bleecker ER, Phillips BR, Mauger DT, Gordon ED, Woodruff PG, Peters MC, Fahy JV; National Heart Lung and Blood Institute (NHLBI) Severe Asthma Research Program (SARP). Mucus plugs in patients with asthma linked to eosinophilia and airflow obstruction. J Clin Invest. 2018 Mar 1;128(3):997-1009. doi: 10.1172/JCI95693. Epub 2018 Feb 5. PMID 29400693
- [Derived] Witt CA, Sheshadri A, Carlstrom L, Tarsi J, Kozlowski J, Wilson B, Gierada DS, Hoffman E, Fain SB, Cook-Granroth J, Sajol G, Sierra O, Giri T, O'Neill M, Zheng J, Schechtman KB, Bacharier LB, Jarjour N, Busse W, Castro M; NHLBI Severe Asthma Research Program (SARP). Longitudinal changes in airway remodeling and air trapping in severe asthma. Acad Radiol. 2014 Aug;21(8):986-93. doi: 10.1016/j.acra.2014.05.001. PMID 25018070
- See also: SARP website — http://www.severeasthma.org